# **Official Title:** Evaluation of Medical Cannabis and Prescription Opioid Taper Support for Reduction of Pain and Opioid Dose in Patients With

Chronic Non-Cancer Pain **NCT Number:** NCT04827992

**Document Date:** 10/22/2024 (MH, CHA Consent)

10/15/2024 (MGH Consent)



General Consent Form Template Version Date: February 2021

| Subject Identification | |
|------------------------|------------------------|
| | Subject Identification |

Protocol Title: Evaluation of Medical Cannabis and Prescription Opioid Taper Support for Reduction of Pain and Opioid Dose in Patients with Chronic Non-cancer Pain

Principal Investigator: Jodi Gilman, PhD

Site Principal Investigator:

Description of Subject Population: Adults with Chronic Non-Cancer Pain on Chronic Opioid Therapy (COT) ages 18-75

#### About this consent form

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

## **Key Information**

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. Your decision won't change the medical care you get within Partners now or in the future.

The following key information is to help you decide whether or not to take part in this research study. We have included more details about the research in the Detailed Information section that follows the key information.

## Why is this research study being done?

In this research study we want to learn more about how medical cannabis may affect opioid use and pain. The goal of this study is for all participants to taper their dose of opioid medications, while managing pain, and receive support from clinicians while doing this through the study





| C1-:4 | . 1.1 4 : 6 4 | |
|---------|---------------|-----|
| Subject | Identificat | ion |

program. Tapering from a medication means gradually reducing your dose. Research has shown that tapering to a reduced dose of opioids may have significant health benefits.

The program is called Prescription Opioid Tapering Support (POTS), which is a behavioral support program aimed at helping you reduce your daily dose of opioid medication.

Everyone in this study will participate in the POTS program, and some people may be able to start using Medical Cannabis (MM) in addition.

### Who will take part in this research?

We are asking you to take part in this study because you are an adult who uses opioid medication to treat your chronic pain.

About 200 people will take part in this study. We plan to enroll participants at Massachusetts General Hospital, Cambridge Health Alliance, and Maine Medical Center.

The National Institute on Drug Abuse is paying for this study to be done.

## How long will you take part in this research study?

If you decide to join this research study, it will take you about 6 months to complete the study. During this time, we will ask you to make 8 study visits to MGH. After the screening visit, we will have you come in for a baseline study visit. You will then come in for visits at 4, 8, 12, 16, 20, and 24 weeks after the baseline visit. The POTS program will take place weekly throughout the study (over 26 weeks).

We will also schedule a call with you one year after your baseline visit to check in on your overall health, medications, and pain levels.

## **Detailed Information**

## What will happen if you take part in this research study?

If you choose to take part in this study, we will ask you to sign this consent form before we do any study procedures.

If you decide to join this research study, we will ask that you:





| Subject | Identificati | on |
|---------|--------------|----|

- Participate in the Prescription Opioid Tapering Support (POTS) program (over 26 weeks)
- Complete questionnaires and participate in interviews asking you about your physical health, mental health, medications, substance use, and overall functioning
- Complete cognitive testing
- Provide urine samples to be tested for THC
- Complete a daily survey about your pain and medications (every day for 28 weeks)
- Confirm scheduled appointments through text message reminders
- If you are of childbearing potential: Agree to use effective contraception (abstinence, hormonal contraception, intra-uterine device, sterilization, or double barrier contraception) during the study.

If you are eligible for this study, you will be randomly assigned to either the active study group (MM+POTS) or a waitlist control group (POTS alone). If you are in the active study group, you will be able to start using medical cannabis right away. If you are in the waitlist control group, you will be asked to abstain from using cannabis, and you will have the option to start using medical cannabis after the first 6 months of the study. Medical marijuana and medical marijuana certificates will not be provided as part of the study.

The POTS program is designed to provide opioid taper support and will be offered weekly to all participants. Sessions will be conducted over videoconference with a trained clinician and other participants. POTS sessions will be focused on individualized problem solving for behavioral self-management of pain and pros and cons of opioid dose taper. POTS sessions will be video recorded. During the 5 regular clinic visits in study weeks 4-20 that coincide with the monthly study visits, study clinicians will work with participants to reduce opioid dose in increments of approximately 10% of the baseline opioid dose. Any opioid dose decrease is optional. Opioid doses will not be increased during the study.

#### Screening Visit:

The purpose of the screening visit is to determine if you are eligible for this study. During your screening visit, we will ask you to:

- Complete several questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Demonstrate how to complete daily surveys on your phone to record your opioid medications and pain levels

#### **Assignment to Study Group**

If after the screening visit, you qualify to take part in this study, we will assign you by chance to the MM group or the control group. You and the study doctor cannot choose your study group.




| Subject Identification |
|------------------------|

We use control groups in research studies to learn if the effects seen in research subjects are truly from a particular treatment.

If you are assigned to the Active Group, you will be able to start using medical cannabis to see if it helps treat your pain or not.

If you are assigned to the Waitlist Group, you will be asked to abstain from cannabis for the first 6 months of the study. If you choose to, you may use cannabis after the 6-month waiting period.

#### **Daily Surveys**

During this study, you will be asked to complete daily surveys to keep track of your marijuana use, opioid use, pain, and health using REDCap, a secure web-based application designed for data collection for research studies.

Study staff will provide instructions for how to access and complete the daily surveys at your screening visit.

You will receive text message reminders containing the survey link when it is time to complete the daily survey. You will be asked to input a four-digit code before completing the survey for your privacy.

This application will NOT be used to collect and report any emergencies, side effects, or adverse events you may experience during the study. If there is something you need to discuss with the site, you should contact study staff directly.

#### **Text Message Reminders**

Text messages by mobile/cell phones are a common form of communication. This research study involves sending you text messages that are relevant to the research study. Texting over mobile/cell phones carries security risks because text messages to mobile/cell phones are not encrypted. This means that information you send or receive by text message could be intercepted or viewed by an unintended recipient, or by your mobile/cell phone provider or carrier.

Below are some important points about texting in this research study.




| Subject Identification |
|------------------------|

- Text messages are not encrypted, and therefore carry security risks. This research study and Mass General Brigham Healthcare are not responsible for any interception of messages sent through unencrypted text message communications.
- You will be responsible for all fees charged by your carrier's service plan for text messaging. This research study and Mass General Brigham Healthcare are not responsible for any increased charges, data usage against plan limits or changes to data fees from the research texts
- Text messaging should not be used in case of an emergency. If you experience a medical emergency, call 911 or go to the nearest hospital emergency department.
- You may decide to not send or receive text messages with staff associated with this research study at any time. You can do this in person or by sending the research number a text message that says, "Stop Research Text."
- Your agreement applies to this research study only. Agreeing to other texts from Mass General Brigham Healthcare, for example appointment reminders, is a separate process. Opting out of other texts from Mass General Brigham Healthcare is a separate process as well.
- It is your responsibility to update your mobile/cell phone number with this research study in the event of a change.

I have had the chance to ask questions about texting with staff associated with this research study. I have been informed of the risks and other information covered above and consent to the use of unencrypted text communications associated with this research study.

| | | <u> </u> |
|---------|------|-----------------|
| Subject | Date | Time (optional) |

#### Baseline Visit:

Approximately, two weeks after your screening visit or once you receive your medical cannabis card if you are in the active group, you will come in for a baseline assessment. During this visit, you will:

- Complete several questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Complete cognitive testing
- Begin the Prescription Opioid Tapering Support (POTS) groups

Visits at (approximately) Weeks 4, 8, 12, 16, 20, and 24:

Approximately, every 4 weeks after the Baseline visit, you will:





| Subject Id | entification |
|------------|--------------|

- Possibly reduce your opioid dose by approximately 10% with consultation with study clinicians
- Complete questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Complete cognitive testing
- Provide a urine sample which will be tested for THC (Visits 2, 4, and 7 only)

#### 12 Month Follow Up Call:

Approximately 12 months after completing your baseline visit, you will complete a follow up call. We will ask you about:

- Your overall health, including physical and mental health
- Your current medications
- Your current substance use

#### Throughout the Study:

Every day of the study (for 28 weeks), you will be asked to complete a short survey on your smartphone/computer asking you about your opioid medication dose and your pain levels.

Every 4 weeks of the study (for weeks 4-24), you will have a study visit (either in person or via zoom), in which you will discuss the possibility of reducing your opioid dose by 10%. You can pause your opioid dose taper at any point. However, you will not be allowed to increase your opioid dose during this study.

We will ask that you tell us about any important changes in your health, even if they do not seem relevant to the research. Partners has an electronic system that lets your study doctors know if you are admitted to a Partners Hospital, or if you visit a Partners Hospital Emergency Department. We want to make sure the study doctors know about any possible problems or side effects you experience while you are taking part in the study.

#### After You Complete the Study:

Study staff will coordinate return to your primary care physician and consult on additional therapy that may help you control your pain and maintain your reduced opioid dose.

#### **Urine Shipments**

We will collect urine samples at three study visits, which will be tested for THC. With your permission, a small quantity (2 teaspoons) of the urine sample will be shipped to collaborators at a lab who can quantify cannabinoids in the urine. We will only ship your sample if a) you agree to having your samples shipped AND b) you report using marijuana products since your last study visit, and/or c) your qualitative urine drug test is positive for THC.





| C 1: (T1 ('C' (' |
|------------------------|
| Subject Identification |

| Do we have your permi | ssion to ship urine | e samples for quantitative analysis? |
|---|---|---|
| YES YES | □ NO | Initials |

#### **Medical Records and Prescription Monitoring Program (PMP)**

This study will require that we access your record through the Prescription Monitoring Program to verify opioid medications and other medications monitored by the PMP.

This study will require that we access your electronic medical record to verify concomitant medications and doses prescribed by caregivers in the MGB, CHA, and MMC systems of care. As part of study procedures, you will provide contact information for your prescribing physician to the study team. The study team will contact the provider(s) primarily responsible for your opioid prescribing at the time of enrollment to inform them of your participation in the study, and again each time you agree to a new opioid dose. Decisions regarding opioid dose adjustment are subject to approval by the prescribing physician.

#### **Information Storage**

Study information collected from you will be stored in a database on a password-protected computer. This information will not become part of your medical record.

We will assign all information a unique code. The key to the code will be kept on encrypted computer. Only the researchers from our research study will be able to use the computer. The code linking test results to subject identity will only be accessible to study staff. If you decide to drop out of this research study at a later time, please contact one of the research coordinators for this study:

- Bryn Evohr: 617-643-4537; bevohr@mgh.harvard.edu
- Julia Jashinski: 617-643-1984; jjashinski@mgh.harvard.edu

## What are the risks and possible discomforts from being in this research study?

Taking part in this research study has some risks that you should consider carefully. Important risks and possible discomforts to know about include:

Reducing opioid dose:





| Subject Identification | |
|------------------------|------------------------|
| Subject Identification | |
| Subject Identification | |
| Subject Identification | |
| Subject Identification | |
| Subject identification | Subject Identification |

Most people don't get very physically uncomfortable with withdrawal while tapering gradually. It is possible you may experience increased pain, restlessness, sweating, body aches, irritability, diarrhea, stomach upset, and sometimes sleep problems.

#### Medical Cannabis:

Cardiovascular effects of cannabis largely depend on several factors, including dose, frequency, route of administration, and duration of use. THC can have diverse effects on heart rate and blood pressure, and although present knowledge about the relationship between cannabis or medical cannabis use and cardiovascular disease outcomes is still limited

Cannabis is associated with reversible effects on appetite, mood, cognition, memory, and perception. At low to moderate doses, THC can produce behavioral intoxication and physiological changes (feeling intoxicated, high, euphoric, dizzy, giddy, tired and lightheaded; increased heart rate, and slowed reaction time). Some participants may experience adverse events including increased anxiety, paranoia, sleeping difficulties, increases in suicidal thoughts, or temporary psychosis. Some people may develop symptoms of cannabis use disorder.

Other risks of medical cannabis may exist that are not known yet. We will inform you of any risks that we learn about as a part of doing this study

#### Loss of confidentiality:

We will not share your identity with anyone outside the Partners/Mass General Brigham institutions. However, we cannot guarantee your total confidentiality.

We will numerically code all data and remove all personal identifiers from the data. We will store all data in password protected databases. Subject information will be accessible only to research staff. Information about study participants will not leave our institution in any form that would identify individual subjects.

## What are possible benefits from being in this research study?

We cannot promise any benefits to you from taking part in this research study. Possible benefits may include reduced opioid dose and better pain management. Others who take opioids for chronic pain may benefit in the future from what we learn in this study.

## What other treatments or procedures are available for your condition?

Other treatments or procedures that are available to treat chronic pain include:

Medications:





| Subject Identification |
|------------------------|

- Over-the-counter medications (acetaminophen, aspirin, ibuprofen, naproxen)
- o Muscle relaxants (cyclobenzaprine, tizanidine, baclofen)
- o Anti-anxiety drugs (lorazepam, diazepam)
- o Antidepressants (amitriptyline, doxepin, imipramine, venlafaxine, duloxetine)
- Prescription anti-inflammatory drugs (celecoxib, piroxicam, indomethacin, meloxicam)
- Other treatments:
  - Steroid injections at the site of pain
  - Surgery
  - Physical and occupational therapy
  - Acupuncture
  - o Massage
  - Hot/cold therapy
  - o Exercise

## If you have questions or concerns about this research study, whom can you call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

Jodi Gilman, Ph.D. is the person in charge of this research study. You can call her at 617-643-7293 Monday through Friday 9AM to 5PM. If necessary, you can reach her after hours at jgilman1@mgh.harvard.edu.

If you have questions about the scheduling of appointments or study visits, please contact one of the research coordinators for this study:

- Bryn Evohr: 617-643-4537; bevohr@mgh.harvard.edu
- Julia Jashinski: 617-643-1984; jjashinski@mgh.harvard.edu

If you want to speak with someone **not** directly involved in this research study, please contact the Mass General Brigham IRB office. You can call them at 857-282-1900.

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure to take part in, or to continue in the research study





| Subject Identification | n |
|------------------------|---|

## How may we use and share your samples and health information for other research?

The information we collect in this study may help advance other research. If you join this study, we remove all information that identifies you (for example, your name, medical record number, and date of birth) and use these de-identified samples and data in other research. It won't be possible to link the information or samples back to you.

## Can you still get medical care within Mass General Brigham if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within Mass General Brigham now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

## What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

## Will you be paid to take part in this research study?

You will be paid following each study visit by check that will be mailed to you. You will earn \$40 for all 8 study visits. You will receive \$30 for completing the 1-Year Phone Call. You will also earn \$20 for each POTS session (26 in total). You will be paid \$1 per day for completing the daily diary and can earn \$10 for full weeks of consecutive entries (up to \$280). You will also be paid up to \$5 per study visit for travel costs. In total, you can earn up to \$1,150 by participating in this study. Regardless of which group you are in (POTS+MM or POTS alone), you can earn the same amount of money. Please see the detailed table here. In accordance with Partners Policy, to receive payment each participant is asked to provide us their Social Security Number or Tax ID number. All payments will be made via check following each study visit. Receiving



General Consent Form Template Version Date: February 2021 Subject Identification

compensation from participating in this study may impact your tax liability and/or eligibility for federal or state benefits (i.e., SSDI, SNAP).

| Week | Visit | | |
|-------|-------------------------------------------------|----|--------|
| -2 | Screening | V0 | \$40 |
| 0 | Baseline | V1 | \$40 |
| 4 | In person | V2 | \$40 |
| 8 | In person | V3 | \$40 |
| 12 | In person | V4 | \$40 |
| 16 | In person | V5 | \$40 |
| 20 | In person | V6 | \$40 |
| 24 | In person | V7 | \$40 |
| 52 | Phone call | | \$30 |
| | Dosing Diaries<br>(28 weeks x<br>\$10/week) | | \$280 |
| | POTS sessions (26<br>sessions x<br>\$20/session | | \$520 |
| Total | | | \$1150 |

## Will I have to pay if I take part in this research study?

There is no cost to you for taking part in this study. The cost of all of the tests and procedures done for research will be paid for by study funds.

You/your health insurer will be responsible for the cost of the MM because this would be needed for your care even if you are not in the study.

Charges for any ongoing or routine medical care you receive outside this study will be billed to you or to your insurance company in the usual way. You will be responsible for any deductibles or co-payments required by your insurer for your routine medical care.




| Subject | Identification | on |
|---------|----------------|----|

# What happens if you are injured as a result of taking part in this research study?

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the beginning of this consent form.

## If you take part in this research study, how will we protect your privacy?

Federal law requires Mass General Brigham to protect the privacy of health information and related information that identifies you. We refer to this information as "identifiable information."

### In this study, we may collect identifiable information about you from:

- Past, present, and future medical records
- Research procedures, including research office visits, tests, interviews, and questionnaires

## Who may see, use, and share your identifiable information and why they may need to do so:

- Mass General Brigham researchers and staff involved in this study
- The sponsor(s) of the study, and people or groups it hires to help perform this research or to audit the research
- Other researchers and medical centers that are part of this study
- The Mass General Brigham ethics board or an ethics board outside Mass General Brigham that oversees the research
- A group that oversees the data (study information) and safety of this study
- Non-research staff within Mass General Brigham who need identifiable information to do their jobs, such as for treatment, payment (billing), or hospital operations (such as assessing the quality of care or research)





| G 1: | . 7.1 .:0 | |
|--------|--------------|------|
| Subjec | t Identifica | tion |

- People or groups that we hire to do certain work for us, such as data storage companies, accreditors, insurers, and lawyers
- Federal agencies (such as the U.S. Department of Health and Human Services (DHHS) and agencies within DHHS like the Food and Drug Administration, the National Institutes of Health, and the Office for Human Research Protections), state agencies, and foreign government bodies that oversee, evaluate, and audit research, which may include inspection of your records
- Public health and safety authorities, if we learn information that could mean harm to you
  or others (such as to make required reports about communicable diseases or about child
  or elder abuse)
- Other:

Some people or groups who get your identifiable information might not have to follow the same privacy rules that we follow and might use or share your identifiable information without your permission in ways that are not described in this form. For example, we understand that the sponsor of this study may use your identifiable information to perform additional research on various products or conditions, to obtain regulatory approval of its products, to propose new products, and to oversee and improve its products' performance. We share your identifiable information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. The sponsor has agreed that it will not contact you without your permission and will not use or share your identifiable information for any mailing or marketing list. However, once your identifiable information is shared outside Mass General Brigham, we cannot control all the ways that others use or share it and cannot promise that it will remain private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your identifiable information. Your permission to use and share your identifiable information does not expire.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifiable information **will not** be used for these purposes without your specific permission.

#### **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your identifiable information for research; however, if you don't sign it, you can't take part in this research study.




| Subject | Identification | on |
|---------|----------------|----|

You have the right to withdraw your permission for us to use or share your identifiable information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study.

You have the right to see and get a copy of your identifiable information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.

#### **Informed Consent and Authorization**

#### **Statement of Person Giving Informed Consent and Authorization**

- I have read this consent form.
- This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study.
- I have had the opportunity to ask questions.
- I understand the information given to me.

#### **Signature of Subject:**

| I give my consent to take part in this research be used and shared as described above. | study and agree to a | llow my health information to |
|---|---|---|
| Subject | Date | Time (optional) |

## **Signature of Study Doctor or Person Obtaining Consent:**

#### **Statement of Study Doctor or Person Obtaining Consent**

• I have explained the research to the study subject.





| on |
|----|

| <ul> <li>I have answered all questions about this</li> </ul> | re answered all questions about this research study to the best of my ability. | |
|---|---|---|
| Study Doctor or Person Obtaining Consent | Date | Time (optional) |

Consent Form Version: 10/10/2024



General Consent Form Template Version Date: February 2021 Subject Identification

Protocol Title: Evaluation of Medical Cannabis and Prescription Opioid Taper Support for Reduction of Pain and Opioid Dose in Patients with Chronic Non-cancer Pain

Principal Investigator: Jodi Gilman, PhD

Site Principal Investigator: Ellie Grossman, MD, MPH

Description of Subject Population: Adults with Chronic Non-Cancer Pain on

Chronic Opioid Therapy (COT) ages 18-75

#### About this consent form

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

## **Key Information**

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. Your decision won't change the medical care you get within Cambridge Health Alliance now or in the future.

The following key information is to help you decide whether or not to take part in this research study. We have included more details about the research in the Detailed Information section that follows the key information.

## Why is this research study being done?

In this research study we want to learn more about how medical cannabis may affect opioid use and pain. The goal of this study is for all participants to taper their dose of opioid medications,





| Subject I | dentifica | ation |
|-----------|-----------|-------|

while managing pain, and receive support from clinicians while doing this through the study program. Tapering from a medication means gradually reducing your dose. Research has shown that tapering to a reduced dose of opioids may have significant health benefits.

The program is called Prescription Opioid Tapering Support (POTS), which is a behavioral support program aimed at helping you reduce your daily dose of opioid medication.

Everyone in this study will participate in the POTS program, and some people may be able to start using Medical Cannabis (MM) in addition.

#### Who will take part in this research?

We are asking you to take part in this study because you are an adult who uses opioid medication to treat your chronic pain.

About 200 people will take part in this study. We plan to enroll participants at Massachusetts General Hospital, Cambridge Health Alliance, and Maine Medical Center.

The National Institute on Drug Abuse is paying for this study to be done.

## How long will you take part in this research study?

If you decide to join this research study, it will take you about 6 months to complete the study. During this time, we will ask you to make 8 study visits to Cambridge Health Alliance (or MGH). After the screening visit, we will have you come in for a baseline study visit. You will then come in for visits at 4, 8, 12, 16, 20, and 24 weeks after the baseline visit. The POTS program will take place weekly throughout the study (over 26 weeks).

We will also schedule a call with you one year after your baseline visit to check in on your overall health, medications, and pain levels.

## **Detailed Information**

## What will happen if you take part in this research study?

If you choose to take part in this study, we will ask you to sign this consent form before we do any study procedures.





| Subject Identification |
|------------------------|

If you decide to join this research study, we will ask that you:

- Participate in the Prescription Opioid Tapering Support (POTS) program (over 26 weeks)
- Complete questionnaires and participate in interviews asking you about your physical health, mental health, medications, substance use, and overall functioning
- Complete cognitive testing
- Provide urine samples to be tested for THC
- Complete a daily survey about your pain and medications (every day for 28 weeks)
- Confirm scheduled appointments through text message reminders
- If you are of childbearing potential: Agree to use effective contraception (abstinence, hormonal contraception, intra-uterine device, sterilization, or double barrier contraception) during the study.

If you are eligible for this study, you will be randomly assigned to either the active study group (MM+POTS) or a waitlist control group (POTS alone). If you are in the active study group, you will be able to start using medical cannabis right away. If you are in the waitlist control group, you will be asked to abstain from using cannabis, and you will have the option to start using medical cannabis after the first 6 months of the study. Medical marijuana and medical marijuana certificates will not be provided as part of the study.

The POTS program is designed to provide opioid taper support and will be offered weekly to all participants. Sessions will be conducted over videoconference with a trained clinician and other participants. POTS sessions will be focused on individualized problem solving for behavioral self-management of pain and pros and cons of opioid dose taper. POTS sessions will be video recorded. During the 5 regular clinic visits in study weeks 4-20 that coincide with the monthly study visits, study clinicians will work with participants to reduce opioid dose in increments of approximately 10% of the baseline opioid dose. Any opioid dose decrease is optional. Opioid doses will not be increased during the study.

#### Screening Visit:

The purpose of the screening visit is to determine if you are eligible for this study. During your screening visit, we will ask you to:

- Complete several questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Demonstrate how to complete daily surveys on your phone to record your opioid medications and pain levels





| Subject Identification |
|------------------------|

#### **Assignment to Study Group**

If after the screening visit, you qualify to take part in this study, we will assign you by chance to the MM group or the control group. You and the study doctor cannot choose your study group.

We use control groups in research studies to learn if the effects seen in research subjects are truly from a particular treatment.

If you are assigned to the Active Group, you will be able to start using medical cannabis to see if it helps treat your pain or not.

If you are assigned to the Waitlist Group, you will be asked to abstain from cannabis for the first 6 months of the study. If you choose to, you may use cannabis after the 6 month waiting period.

#### **Daily Surveys**

During this study, you will be asked to complete daily surveys to keep track of your marijuana use, opioid use, pain, and health using REDCap, a secure web-based application designed for data collection for research studies.

Study staff will provide instructions for how to access and complete the daily surveys at your screening visit.

You will receive text message reminders containing the survey link when it is time to complete the daily survey. You will be asked to input a four-digit code before completing the survey for your privacy.

This application will NOT be used to collect and report any emergencies, side effects, or adverse events you may experience during the study. If there is something you need to discuss with the site, you should contact study staff directly.

#### **Text Message Reminders**

Text messages by mobile/cell phones are a common form of communication. This research study involves sending you text messages that are relevant to the research study. Texting over mobile/cell phones carries security risks because text messages to mobile/cell phones are not encrypted. This means that information you send or receive by text message could be intercepted or viewed by an unintended recipient, or by your mobile/cell phone provider or carrier.




| Subject Identification |
|------------------------|

Below are some important points about texting in this research study.

- Text messages are not encrypted, and therefore carry security risks. This research study and Mass General Brigham Healthcare are not responsible for any interception of messages sent through unencrypted text message communications.
- You will be responsible for all fees charged by your carrier's service plan for text messaging. This research study and Mass General Brigham Healthcare are not responsible for any increased charges, data usage against plan limits or changes to data fees from the research texts
- Text messaging should not be used in case of an emergency. If you experience a medical emergency, call 911 or go to the nearest hospital emergency department.
- You may decide to not send or receive text messages with staff associated with this research study at any time. You can do this in person or by sending the research number a text message that says, "Stop Research Text."
- Your agreement applies to this research study only. Agreeing to other texts from Mass General Brigham Healthcare, for example appointment reminders, is a separate process. Opting out of other texts from Mass General Brigham Healthcare is a separate process as well.
- It is your responsibility to update your mobile/cell phone number with this research study in the event of a change.

I have had the chance to ask questions about texting with staff associated with this research study. I have been informed of the risks and other information covered above and consent to the use of unencrypted text communications associated with this research study.

| Subject | Date | Time (optional) |
|---------|------|-----------------|

#### Baseline Visit:

Approximately, two weeks after your screening visit or once you receive your medical cannabis card if you are in the active group, you will come in for a baseline assessment. During this visit, you will:

- Complete several questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Complete cognitive testing
- Begin the Prescription Opioid Tapering Support (POTS) groups

Visits at (approximately) Weeks 4, 8, 12, 16, 20, and 24:





| Subject Identification |
|------------------------|

Approximately, every 4 weeks after the Baseline visit, you will:

- Possibly reduce your opioid dose by approximately 10% with consultation with study clinicians
- Complete questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Complete cognitive testing
- Provide a urine sample which will be tested for THC (Visits 2, 4, and 7 only)

#### 12 Month Follow Up Call:

Approximately 12 months after completing your baseline visit, you will complete a follow up call. We will ask you about:

- Your overall health, including physical and mental health
- Your current medications
- Your current substance use

#### Throughout the Study:

Every day of the study (for 28 weeks), you will be asked to complete a short survey on your smartphone/computer asking you about your opioid medication dose and your pain levels.

Every 4 weeks of the study (for weeks 4-24), you will have a study visit (either in person or via zoom), in which you will discuss the possibility of reducing your opioid dose by 10%. You can pause your opioid dose taper at any point. However, you will not be allowed to increase your opioid dose during this study.

We will ask that you tell us about any important changes in your health, even if they do not seem relevant to the research. MGB has an electronic system that lets your study doctors know if you are admitted to a MGB Hospital, or if you visit an MGB Emergency Department. We want to make sure the study doctors know about any possible problems or side effects you experience while you are taking part in the study.

#### After You Complete the Study:

Study staff will coordinate return to your primary care physician and consult on additional therapy that may help you control your pain and maintain your reduced opioid dose.

#### **Urine Shipments**

We will collect urine samples at three study visits, which will be tested for THC. With your permission, a small quantity (2 teaspoons) of the urine sample will be shipped to collaborators at a lab who can quantify cannabinoids in the urine. We will only ship your sample if a) you agree





| Subject Identification |
|------------------------|

to having your samples shipped AND b) you report using marijuana products since your last study visit, and/or c) your qualitative urine drug test is positive for THC.

| Do we have your permissi | ion to ship urine | samples for quantitative analysis? |
|---|---|---|
| <b>YES</b> | □ NO | Initials |

#### **Medical Records and Prescription Monitoring Program (PMP)**

This study will require that we access your record through the Prescription Monitoring Program to verify opioid medications and other medications monitored by the PMP.

This study will require that we access your electronic medical record to verify concomitant medications and doses prescribed by caregivers in the MGB, CHA, and MMC systems of care. As part of study procedures, you will provide contact information for your prescribing physician to the study team. The study team will contact the provider(s) primarily responsible for your opioid prescribing at the time of enrollment to inform them of your participation in the study, and again each time you agree to a new opioid dose. Decisions regarding opioid dose adjustment are subject to approval by the prescribing physician.

#### **Information Storage**

Study information collected from you will be stored in a database on a password-protected computer. This information will not become part of your medical record.

We will assign all information a unique code. The key to the code will be kept on encrypted computer. Only the researchers from our research study will be able to use the computer. The code linking test results to subject identity will only be accessible to study staff. If you decide to drop out of this research study at a later time, please contact one of the research coordinators for this study:

Unity Ikeasoguh: 781-605-5005; nikeasoguh@challiance.org

# What are the risks and possible discomforts from being in this research study?

Taking part in this research study has some risks that you should consider carefully. Important risks and possible discomforts to know about include:





| Subject Identification |
|------------------------|

#### Reducing opioid dose:

Most people don't get very physically uncomfortable with withdrawal while tapering gradually. It is possible you may experience increased pain, restlessness, sweating, body aches, irritability, diarrhea, stomach upset, and sometimes sleep problems.

#### Medical Cannabis:

Cardiovascular effects of cannabis largely depend on several factors, including dose, frequency, route of administration, and duration of use. THC can have diverse effects on heart rate and blood pressure, and although present knowledge about the relationship between cannabis or medical cannabis use and cardiovascular disease outcomes is still limited

Cannabis is associated with reversible effects on appetite, mood, cognition, memory, and perception. At low to moderate doses, THC can produce behavioral intoxication and physiological changes (feeling intoxicated, high, euphoric, dizzy, giddy, tired and lightheaded; increased heart rate, and slowed reaction time). Some participants may experience adverse events including increased anxiety, paranoia, sleeping difficulties, increases in suicidal thoughts or temporary psychosis. Some people may develop symptoms of cannabis use disorder.

Other risks of medical cannabis may exist that are not known yet. We will inform you of any risks that we learn about as a part of doing this study

#### Loss of confidentiality:

We will not share your identity with anyone outside the Cambridge Health Alliance and Mass General Brigham institutions. However, we cannot guarantee your total confidentiality.

We will numerically code all data and remove all personal identifiers from the data. We will store all data in password protected databases. Subject information will be accessible only to research staff. Information about study participants will not leave our institution in any form that would identify individual subjects.

## What are possible benefits from being in this research study?

We cannot promise any benefits to you from taking part in this research study. Possible benefits may include reduced opioid dose and better pain management. Others who take opioids for chronic pain may benefit in the future from what we learn in this study.

What other treatments or procedures are available for your condition?





| Subject Ident | · c· .· |
|---------------|-------------|

Other treatments or procedures that are available to treat chronic pain include:

- Medications:
  - Over-the-counter medications (acetaminophen, aspirin, ibuprofen, naproxen)
  - o Muscle relaxants (cyclobenzaprine, tizanidine, baclofen)
  - Anti-anxiety drugs (lorazepam, diazepam)
  - o Antidepressants (amitriptyline, doxepin, imipramine, venlafaxine, duloxetine)
  - Prescription anti-inflammatory drugs (celecoxib, piroxicam, indomethacin, meloxicam)
- Other treatments:
  - o Steroid injections at the site of pain
  - Surgery
  - Physical and occupational therapy
  - o Acupuncture
  - o Massage
  - Hot/cold therapy
  - o Exercise

## If you have questions or concerns about this research study, whom can you call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

Jodi Gilman, Ph.D. is the person in charge of this research study. You can call her at 617-643-7293 Monday through Friday 9AM to 5PM. If necessary, you can reach her after hours at <a href="mailto:jgilman1@mgh.harvard.edu">jgilman1@mgh.harvard.edu</a>.

Ellie Grossman, MD, MPH is the person in charge of this study at Cambridge Health Alliance. You can call her at 617-591-6300 Monday through Friday 8am to 5pm, and there is an afterhours on-call service for urgent situations.

If you have questions about the scheduling of appointments or study visits, please contact one of the research coordinators for this study:

Unity Ikeasoguh: 781-605-5005; nikeasoguh@challiance.org







If you want to speak with someone **not** directly involved in this research study, please contact the Mass General Brigham IRB office. You can call them at 857-282-1900.

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure to take part in, or to continue in the research study

## How may we use and share your samples and health information for other research?

The information we collect in this study may help advance other research. If you join this study, we remove all information that identifies you (for example, your name, medical record number, and date of birth) and use these de-identified samples and data in other research. It won't be possible to link the information or samples back to you.

# Can you still get medical care within Cambridge Health Alliance if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within Cambridge Health Alliance now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

## What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

## Will you be paid to take part in this research study?




General Consent Form Template Version Date: February 2021 Subject Identification

You will be paid following each study visit by check that will be mailed to you. You will earn \$40 for all 8 study visits. You will receive \$30 for completing the 1-Year Phone Call. You will also earn \$20 for each POTS session (26 in total). You will be paid \$1 per day for completing the daily diary and can earn \$10 for full weeks of consecutive entries (up to \$280). You will also be paid up to \$5 per study visit for travel costs. In total, you can earn up to \$1,150 by participating in this study. Regardless of which group you are in (POTS+MM or POTS alone), you can earn the same amount of money. Please see the detailed table here. In accordance with MGB Policy, to receive payment each participant is asked to provide us their Social Security Number or Tax ID number. All payments will be made via check following each study visit. Receiving compensation from participating in this study may impact your tax liability and/or eligibility for federal or state benefits (i.e., SSDI, SNAP).

| Week | Visit | | |
|-------|---------------------------------------------|----|--------|
| -2 | Screening | V0 | \$40 |
| 0 | Baseline | V1 | \$40 |
| 4 | In person | V2 | \$40 |
| 8 | In person | V3 | \$40 |
| 12 | In person | V4 | \$40 |
| 16 | In person | V5 | \$40 |
| 20 | In person | V6 | \$40 |
| 24 | In person | V7 | \$40 |
| 52 | Phone call | | \$30 |
| | Dosing Diaries<br>(28 weeks x<br>\$10/week) | | \$280 |
| | POTS sessions (26 | | |
| | sessions x | | \$520 |
| | \$20/session | | |
| Total | | | \$1150 |

## Will I have to pay if I take part in this research study?

There is no cost to you for taking part in this study. The cost of all of the tests and procedures done for research will be paid for by study funds.





| Subject Identification |
|------------------------|

You/your health insurer will be responsible for the cost of the MM because this would be needed for your care even if you are not in the study.

Charges for any ongoing or routine medical care you receive outside this study will be billed to you or to your insurance company in the usual way. You will be responsible for any deductibles or co-payments required by your insurer for your routine medical care.

## What happens if you are injured as a result of taking part in this research study?

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the beginning of this consent form.

## If you take part in this research study, how will we protect your privacy?

Federal law requires Mass General Brigham to protect the privacy of health information and related information that identifies you. We refer to this information as "identifiable information."

## In this study, we may collect identifiable information about you from:

- Past, present, and future medical records
- Research procedures, including research office visits, tests, interviews, and questionnaires

## Who may see, use, and share your identifiable information and why they may need to do so:

- Mass General Brigham researchers and staff involved in this study
- Cambridge Health Alliance researchers and staff involved in this study







- The sponsor(s) of the study, and people or groups it hires to help perform this research or to audit the research
- Other researchers and medical centers that are part of this study
- The Mass General Brigham ethics board or an ethics board outside Mass General Brigham that oversees the research
- A group that oversees the data (study information) and safety of this study
- Non-research staff within Mass General Brigham who need identifiable information to do their jobs, such as for treatment, payment (billing), or hospital operations (such as assessing the quality of care or research)
- People or groups that we hire to do certain work for us, such as data storage companies, accreditors, insurers, and lawyers
- Federal agencies (such as the U.S. Department of Health and Human Services (DHHS) and agencies within DHHS like the Food and Drug Administration, the National Institutes of Health, and the Office for Human Research Protections), state agencies, and foreign government bodies that oversee, evaluate, and audit research, which may include inspection of your records
- Public health and safety authorities, if we learn information that could mean harm to you or others (such as to make required reports about communicable diseases or about child or elder abuse)
- Other:

Some people or groups who get your identifiable information might not have to follow the same privacy rules that we follow and might use or share your identifiable information without your permission in ways that are not described in this form. We share your identifiable information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. However, once your identifiable information is shared outside Mass General Brigham, we cannot control all the ways that others use or share it and cannot promise that it will remain private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your identifiable information. Your permission to use and share your identifiable information does not expire.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifiable information **will not** be used for these purposes without your specific permission.





| Subject Identification |
|------------------------|

#### **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your identifiable information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your identifiable information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study.

You have the right to see and get a copy of your identifiable information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.

#### **Informed Consent and Authorization**

#### **Statement of Person Giving Informed Consent and Authorization**

- I have read this consent form.
- This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study.
- I have had the opportunity to ask questions.
- I understand the information given to me.

#### Signature of Subject:

| | n this research study and agree to allo | ow my health information to |
|---|---|---|
| be used and shared as described | l above. | |
| Subject | Date | Time (optional) |
| | D 14 . £15 | |





| Subject Identification |
|------------------------|

### **Signature of Study Doctor or Person Obtaining Consent:**

### **Statement of Study Doctor or Person Obtaining Consent**

- I have explained the research to the study subject.
- I have answered all questions about this research study to the best of my ability.

Study Doctor or Person Obtaining Consent Date Time (optional)

Consent Form Version: 10/18/2024




| Subject Identification |
|------------------------|

Protocol Title: Evaluation of Medical Cannabis and Prescription Opioid Taper Support for Reduction of Pain and Opioid Dose in Patients with Chronic

Non-cancer Pain

Principal Investigator: Jodi Gilman, PhD

Site Principal Investigator: Aurora Quaye, MD

Description of Subject Population: Adults with Chronic Non-Cancer Pain on

Chronic Opioid Therapy (COT) ages 18-75

#### About this consent form

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

## **Key Information**

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. Your decision won't change the medical care you get within MaineHealth now or in the future.

The following key information is to help you decide whether or not to take part in this research study. We have included more details about the research in the Detailed Information section that follows the key information.

## Why is this research study being done?

In this research study we want to learn more about how medical cannabis may affect opioid use and pain. The goal of this study is for all participants to taper their dose of opioid medications, while managing pain, and receive support from clinicians while doing this through the study





| l | |
|---|------------------------|
| l | |
| l | |
| | Subject Identification |

program. Tapering from a medication means gradually reducing your dose. Research has shown that tapering to a reduced dose of opioids may have significant health benefits.

The program is called Prescription Opioid Tapering Support (POTS), which is a behavioral support program aimed at helping you reduce your daily dose of opioid medication.

Everyone in this study will participate in the POTS program, and some people may be able to start using Medical Cannabis (MM) in addition.

### Who will take part in this research?

We are asking you to take part in this study because you are an adult who uses opioid medication to treat your chronic pain.

About 200 people will take part in this study. We plan to enroll participants at Massachusetts General Hospital (MGH), Cambridge Health Alliance (CHA), and MaineHealth (MMC).

The National Institute on Drug Abuse is paying for this study to be done.

## How long will you take part in this research study?

If you decide to join this research study, it will take you about 6 months to complete the study. During this time, we will ask you to make 8 study visits through MaineHealth. After the screening visit, we will have you come in for a baseline study visit. You will then come in for visits at 4, 8, 12, 16, 20, and 24 weeks after the baseline visit. The POTS program will take place weekly throughout the study (over 26 weeks).

We will also schedule a call with you one year after your baseline visit to check in on your overall health, medications, and pain levels.

#### What are the most common risks and the most serious risks?

#### Risks of reducing opioid dose:

Most people don't get very physically uncomfortable with withdrawal while tapering gradually. It is possible you may experience increased pain, restlessness, sweating, body aches, irritability, diarrhea, stomach upset, and sometimes sleep problems.

Risks of using Medical Cannabis:







Some participants may experience adverse events including increased anxiety, paranoia, sleeping difficulties, increases in suicidal thoughts or temporary psychosis. Some people may develop symptoms of cannabis use disorder.

## **Detailed Information**

## What will happen if you take part in this research study?

If you choose to take part in this study, we will ask you to sign this consent form before we do any study procedures.

If you decide to join this research study, we will ask that you:

- Participate in the Prescription Opioid Tapering Support (POTS) program (over 26 weeks)
- Complete questionnaires and participate in interviews asking you about your physical health, mental health, medications, substance use, and overall functioning
- Complete cognitive testing
- Provide urine samples to be tested for THC
- Complete a daily survey about your pain and medications (every day for 28 weeks)
- Confirm scheduled appointments through text message reminders
- If you are of childbearing potential: Agree to use effective contraception (abstinence, hormonal contraception, intra-uterine device, sterilization, or double barrier contraception) during the study.

If you are eligible for this study, you will be randomly assigned to either the active study group (MM+POTS) or a waitlist control group (POTS alone). If you are in the active study group, you will be able to start using medical cannabis right away. If you are in the waitlist control group, you will be asked to abstain from using cannabis, and you will have the option to start using medical cannabis after the first 6 months of the study. Medical marijuana and medical marijuana certificates will not be provided as part of the study.

The POTS program is designed to provide opioid taper support and will be offered weekly to all participants. Sessions will be conducted over videoconference with a trained clinician and other participants. POTS sessions will be focused on individualized problem solving for behavioral self-management of pain and pros and cons of opioid dose taper. POTS sessions will be video recorded. During the 5 regular clinic visits in study weeks 4-20 that coincide with the monthly study visits, study clinicians will work with participants to reduce opioid dose in increments of approximately 10% of the baseline opioid dose. Any opioid dose decrease is optional. Opioid





| Subject Identification |
|------------------------|

doses will not be increased during the study.




| Subject Identification |
|------------------------|

#### Screening Visit:

The purpose of the screening visit is to determine if you are eligible for this study. During your screening visit, we will ask you to:

- Complete several questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Demonstrate how to complete daily surveys on your phone to record your opioid medications and pain levels

#### **Assignment to Study Group**

If after the screening visit, you qualify to take part in this study, we will assign you by chance to the MM group or the control group. You and the study doctor cannot choose your study group.

We use control groups in research studies to learn if the effects seen in research subjects are truly from a particular treatment.

If you are assigned to the Active Group, you will be able to start using medical cannabis to see if it helps treat your pain or not.

If you are assigned to the Waitlist Group, you will be asked to abstain from cannabis for the first 6 months of the study. If you choose to, you may use cannabis after the 6 month waiting period.

#### **Daily Surveys**

During this study, you will be asked to complete daily surveys to keep track of your marijuana use, opioid use, pain, and health using REDCap, a secure web-based application designed for data collection for research studies.

Study staff will provide instructions for how to access and complete the daily surveys at your screening visit.

You will receive text message reminders containing the survey link when it is time to complete the daily survey. You will be asked to input a four-digit code before completing the survey for your privacy.

This application will NOT be used to collect and report any emergencies, side effects, or adverse events you may experience during the study. If there is something you need to discuss with the site, you should contact study staff directly.




| Subject Identification |
|------------------------|

#### **Text Message Reminders**

Text messages by mobile/cell phones are a common form of communication. This research study involves sending you text messages that are relevant to the research study. Texting over mobile/cell phones carries security risks because text messages to mobile/cell phones are not encrypted. This means that information you send or receive by text message could be intercepted or viewed by an unintended recipient, or by your mobile/cell phone provider or carrier.

Below are some important points about texting in this research study.

- Text messages are not encrypted, and therefore carry security risks. This research study, Mass General Brigham Healthcare and MaineHealth are not responsible for any interception of messages sent through unencrypted text message communications.
- You will be responsible for all fees charged by your carrier's service plan for text
  messaging. This research study, Mass General Brigham Healthcare and MaineHealth are
  not responsible for any increased charges, data usage against plan limits or changes to
  data fees from the research texts
- Text messaging should not be used in case of an emergency. If you experience a medical emergency, call 911 or go to the nearest hospital emergency department.
- You may decide to not send or receive text messages with staff associated with this research study at any time. You can do this in person or by sending the research number a text message that says, "Stop Research Text."
- Your agreement applies to this research study only. Agreeing to other texts from Mass General Brigham Healthcare and MaineHealth, for example appointment reminders, is a separate process. Opting out of other texts from Mass General Brigham Healthcare and MaineHealth is a separate process as well.
- It is your responsibility to update your mobile/cell phone number with this research study in the event of a change.

I have had the chance to ask questions about texting with staff associated with this research study. I have been informed of the risks and other information covered above and consent to the use of unencrypted text communications associated with this research study.

| use of unenerypted text communications associated with this research study. | | |
|---|---|---|
| Subject | Date | Time (optional) |
| Baseline Visit: | | |







Approximately, two weeks after your screening visit or once you receive your medical cannabis card if you are in the active group, you will come in for a baseline assessment. During this visit, you will:

- Complete several questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Complete cognitive testing
- Begin the Prescription Opioid Tapering Support (POTS) groups

#### <u>Visits at (approximately) Weeks 4, 8, 12, 16, 20, and 24:</u>

Approximately, every 4 weeks after the Baseline visit, you will:

- Possibly reduce your opioid dose by approximately 10% with consultation with study clinicians
- Complete questionnaires
- Participate in interviews asking about physical health, mental health, and substance use
- Complete cognitive testing
- Provide a urine sample which will be tested for THC (Visits 2, 4, and 7 only)

#### 12 Month Follow Up Call:

Approximately 12 months after completing your baseline visit, you will complete a follow up call. We will ask you about:

- Your overall health, including physical and mental health
- Your current medications
- Your current substance use

#### Throughout the Study:

Every day of the study (for 28 weeks), you will be asked to complete a short survey on your smartphone/computer asking you about your opioid medication dose and your pain levels.

Every 4 weeks of the study (for weeks 4-24), you will have a study visit (either in person or via zoom), in which you will discuss the possibility of reducing your opioid dose by 10%. You can pause your opioid dose taper at any point. However, you will not be allowed to increase your opioid dose during this study.

We will ask that you tell us about any important changes in your health, even if they do not seem relevant to the research. We want to make sure the study doctors know about any possible problems or side effects you experience while you are taking part in the study.

After You Complete the Study:





| Subject Identification |
|------------------------|

Study staff will coordinate return to your primary care physician and consult on additional therapy that may help you control your pain and maintain your reduced opioid dose.

#### **Urine Shipments**

We will collect urine samples at three study visits, which will be tested for THC. With your permission, a small quantity (2 teaspoons) of the urine sample will be shipped to collaborators at a lab who can quantify cannabinoids in the urine. We will only ship your sample if a) you agree to having your samples shipped AND b) you report using marijuana products since your last study visit, and/or c) your qualitative urine drug test is positive for THC.

| Do we have your permission to ship urine samples for quantitative analysis? | | |
|---|---|---|
| <b>YES</b> | □ NO | Initials |

#### Medical Records and Prescription Monitoring Program (PMP)

This study will require that we access your record through the Prescription Monitoring Program to verify opioid medications and other medications monitored by the PMP.

This study will require that we access your electronic medical record to verify concomitant medications and doses prescribed by caregivers in the MGB, CHA, and MMC systems of care. As part of study procedures, you will provide contact information for your prescribing physician to the study team. The study team will contact the provider(s) primarily responsible for your opioid prescribing at the time of enrollment to inform them of your participation in the study, and again each time you agree to a new opioid dose. Decisions regarding opioid dose adjustment are subject to approval by the prescribing physician.

#### **Information Storage**

Study information collected from you will be stored in a database on a password-protected computer at Massachusetts General Brigham. This information will not become part of your medical record.

They will assign all information a unique code. The key to the code will be kept on encrypted computer. Only the researchers from our research study will be able to use the computer. The code linking test results to subject identity will only be accessible to study staff. If you decide todrop out of this research study at a later time, please contact one of the research coordinators forthis study. Anna Cloutier, RN, BSN - 207-396-8304 email: anna.cloutier@mainehealth.org





| Subject Identification |
|------------------------|

# What are the risks and possible discomforts from being in this research study?

Taking part in this research study has some risks that you should consider carefully. Important risks and possible discomforts to know about include:

#### Reducing opioid dose:

Most people don't get very physically uncomfortable with withdrawal while tapering gradually. It is possible you may experience increased pain, restlessness, sweating, body aches, irritability, diarrhea, stomach upset, and sometimes sleep problems.

#### Medical Cannabis:

Cardiovascular effects of cannabis largely depend on several factors, including dose, frequency, route of administration, and duration of use. THC can have diverse effects on heart rate and blood pressure, and although present knowledge about the relationship between cannabis or medical cannabis use and cardiovascular disease outcomes is still limited

Cannabis is associated with reversible effects on appetite, mood, cognition, memory, and perception. At low to moderate doses, THC can produce behavioral intoxication and physiological changes (feeling intoxicated, high, euphoric, dizzy, giddy, tired and lightheaded; increased heart rate, and slowed reaction time). Some participants may experience adverse events including increased anxiety, paranoia, sleeping difficulties, increases in suicidal thoughts or temporary psychosis. Some people may develop symptoms of cannabis use disorder.

Other risks of medical cannabis may exist that are not known yet. We will inform you of any risks that we learn about as a part of doing this study

#### Loss of confidentiality:

We will not share your identity with anyone outside the Partners/Mass General Brigham and MaineHealth institutions. However, we cannot guarantee your total confidentiality.

We will numerically code all data and remove all personal identifiers from the data. We will store all data in password protected databases. Subject information will be accessible only to research staff. Information about study participants will not leave our institution in any form that would identify individual subjects.




| Subject Identification |
|------------------------|

## What are possible benefits from being in this research study?

We cannot promise any benefits to you from taking part in this research study. Possible benefits may include reduced opioid dose and better pain management. Others who take opioids for chronic pain may benefit in the future from what we learn in this study.

## What other treatments or procedures are available for your condition?

Other treatments or procedures that are available to treat chronic pain include:

- Medications:
  - Over-the-counter medications (acetaminophen, aspirin, ibuprofen, naproxen)
  - o Muscle relaxants (cyclobenzaprine, tizanidine, baclofen)
  - o Anti-anxiety drugs (lorazepam, diazepam)
  - o Antidepressants (amitriptyline, doxepin, imipramine, venlafaxine, duloxetine)
  - Prescription anti-inflammatory drugs (celecoxib, piroxicam, indomethacin, meloxicam)
- Other treatments:
  - Steroid injections at the site of pain
  - Surgery
  - Physical and occupational therapy
  - o Acupuncture
  - o Massage
  - Hot/cold therapy
  - Exercise

## If you have questions or concerns about this research study, whom can you call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

<u>Aurora Quaye, MD</u> is the person in charge of this research study at MaineHealth. You can call her at <u>207-200-4061</u> at any time during your enrollment in the study.

If you have questions about the scheduling of appointments or study visits, please contact the research coordinator for this study:

**Anna Cloutier at 207-396-8304** 





| Subject Identification |
|------------------------|

Jodi Gilman, Ph.D. is the person in charge of this research study. You can call her at 617-643-7293 Monday through Friday 9AM to 5PM. If necessary, you can reach her after hours at jgilman1@mgh.harvard.edu.

If you want to speak with someone **not** directly involved in this research study, please contact the <u>Mass General Brigham IRB</u> office. You can call them at 857-282-1900.

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure to take part in, or to continue in the research study

## How may we use and share your samples and health information for other research?

The information we collect in this study may help advance other research. If you join this study, we remove all information that identifies you (for example, your name, medical record number, and date of birth) and use these de-identified samples and data in other research. It won't be possible to link the information or samples back to you.

## Can you still get medical care within MaineHealth if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within MaineHealth now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

## What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

If you want to withdraw, please contact the study Principal Investigator or the Research 






Coordinator, Anna Cloutier, at: 207-396-8304. She will answer any questions that you have and will help you to stop the study safely.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. Ifthis happens, we will tell you why. We will also help arrange other care for you, if needed.

### Will you be paid to take part in this research study?

You will be paid following each study visit by check that will be mailed to you. You will earn \$40 for all 8 study visits. You will receive \$30 for completing the 1-Year Phone Call. You will also earn \$20 for each POTS session(26 in total). You will be paid \$1 per day for completing the daily diary and can earn \$10 for fullweeks of consecutive entries (up to \$280). You will also be paid up to \$5 per study visit for travel costs. In total, you can earn up to \$1,150 by participating in this study. Regardless of which group you are in (POTS+MM or POTS alone), you can earn the same amount of money. Please see the detailed table here. In accordance with Partners Policy, to receive payment each participant is asked to provide us their Social Security Number or Tax ID number. All payments will be made via check following each study visit. Receiving compensation from participating inthis study may impact your tax liability and/or eligibility for federal or state benefits (i.e., SSDI, SNAP).

| Week | Visit | | |
|-------|-------------------------------------------------|----|--------|
| -2 | Screening | V0 | \$40 |
| 0 | Baseline | V1 | \$40 |
| 4 | In person | V2 | \$40 |
| 8 | In person | V3 | \$40 |
| 12 | In person | V4 | \$40 |
| 16 | In person | V5 | \$40 |
| 20 | In person | V6 | \$40 |
| 24 | In person | V7 | \$40 |
| 52 | Phone call | | \$30 |
| | Dosing Diaries<br>(28 weeks x<br>\$10/week) | | \$280 |
| | POTS sessions (26<br>sessions x<br>\$20/session | | \$520 |
| Total | | | \$1150 |







## Will I have to pay if I take part in this research study?

There is no cost to you for taking part in this study. The cost of all of the tests and procedures done for research will be paid for by study funds.

This study will not pay for or supply the MM that you use for pain management and you/your health insurer will be responsible for the cost of the MM.

Charges for any ongoing or routine medical care you receive outside this study will be billed to you or to your insurance company in the usual way. You will be responsible for any deductibles or co-payments required by your insurer for your routine medical care.

# What happens if you are injured as a result of taking part in this research study?

In the case of injury or illness resulting from this research study, medical treatment will be available at the usual charge.

MaineHealth has no policy or plan to pay for any injuries that you might receive as a result of your participation in this study. However, this does not take away your rights to seek or collect compensation for injury related to malpractice, fault, or blame on the part of those involved in the research, including the hospital.

You or your insurance company will be responsible for any costs resulting from underlying disease or treatments provided to you outside of this research study.




| Subject Identification |
|------------------------|

## Permission for the research team to obtain and use your patient health information

### How will the privacy of my patient health information be protected?

There are state and federal privacy laws that protect the use and sharing of your patient health information. By signing this form, you provide your permission, called your "authorization," for the use and sharing of patient health information protected by the Privacy Rule. Authorization includes allowing:

- Your health care providers to share your health information for this research study
- The research team to use and share your health information for this research study.

Health information about you that will be used or shared with others involved in this study may include your research record and any health care records at MaineHealth. Specifically, this will include: your name, date of birth, medical record number, phone number, email address, mailing address, social security number (for payment purposes), and dates of past medical events. This may also include any new health information about you that comes from the research tests or procedures described in this consent form. Psychotherapy notes in your health records (if any) will not, however, be shared or used. Use of these notes requires a separate, signed authorization.

The research team and people within MaineHealth who oversee and help administer research may see, use or share your information as needed for the research.

People outside of MaineHealth may need to see or receive your information for this study. Specifically, Massachusetts General Hospital. Other examples include government agencies (such as the Food and Drug Administration), safety monitors, other sites in the study and companies that sponsor the study.

We cannot do this study without your authorization to use and share your information. You do not have to give us this authorization. If you do not, then you may not join this study.

We will use and share your information only as described in this form; however, people outside MaineHealth who receive your information may not be covered by this promise or by the federal Privacy Rule. We try to make sure that everyone who needs to see your information keeps it confidential – but we cannot guarantee that your information will not be re-disclosed.







The use and sharing of your information has no time limit. You may revoke (cancel) your permission to use and share your information at any time by notifying the Principal Investigator of this study by phone or in writing. If you contact the Principal Investigator by phone, you must follow-up with a written request that includes the study number and your contact information. Send your request to: *Dr. Aurora Quaye*, 81 Research Drive, Scarborough, ME 04074; Attn: Anna Cloutier, RN, CTO.

If you do cancel your authorization to use and share your information, your part in this study will end and no further information about you will be collected. Your revocation (cancellation) would not affect information already collected in the study, or information we shared before you wrote to the Principal Investigator to cancel your authorization.

Your decision to not sign this authorization will not affect any other treatment, health care, enrollment in health plans or eligibility for benefits.

Signing this authorization also means that you will not be able to see or copy your study-related information until the study is completed. This includes any portion of your medical records that describes study treatment.

Finally, with your initials, please specifically authorize the use of your private health information relating substance abuse, mental health information, or HIV/AIDS, if applicable, for the above-described purposes.

| Initia | als: |
|---------|------|
| 1111111 | ars. |

#### **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your identifiable information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your identifiable information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study.




You have the right to see and get a copy of your identifiable information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.

### **Informed Consent and Authorization**

### **Statement of Person Giving Informed Consent and Authorization**

- I have read this consent form.
- This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study.

to

- I have had the opportunity to ask questions.
- I understand the information given to me.

### **Signature of Subject:**

| I give my consent to take part in this research st<br>be used and shared as described above. | tudy and agree to a | llow my health information |
|---|---|---|
| Subject | Date | Time (optional) |
| Signature of Study Doctor or Person C | Obtaining Cons | ent: |
| Statement of Study Doctor or Person Obtain | ing Consent | |
| <ul> <li>I have explained the research to the stud</li> <li>I have answered all questions about this</li> </ul> | • | the best of my ability. |
| Study Doctor or Person Obtaining Consent | Date | Time (optional) |
| Consent Form Version: 10/18/2024 | | |

